CLINICAL TRIAL: NCT03247361
Title: The Addition of High-intensity vs. Low-intensity Inspiratory Muscle Training to Combined Aerobic and Resistance Exercise in Patients With Heart Failure
Brief Title: High-intensity vs. Low-intensity Inspiratory Muscle Training in Patients With Heart Failure
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Federal University of Bahia (Other)
Responsible Party: Principal Investigator, Mansueto Gomes Neto, Principal researcher, Federal University of Bahia
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: FUBahia HIIT IMT
Record Dates: First submitted 2017-08-09; First posted 2017-08-11 (Actual); Last update posted 2018-11-07 (Actual); Status verified 2018-11

CONDITIONS: Heart Failure
Keywords: Heart Failure; Rehabilitation
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- High-intensity IMT (Experimental): High-intensity IMT + Aerobic/resistance exercise
  IMT: Training loads will be adjusted weekly to the maximal inspiratory pressure (MIP). In the first 2 weeks as adaptation, the protocol will be of 2 minutes warm-up with intensity 20% of MIP. The training will have 7 peaks of intensity with 70% of MIP for 30 sec, with 30-sec of passive rest between the peaks, finishing the training with 20% of MIP for 2 min, totaling 10 min and 30 sec. From the third week the protocol will be of 2 min warm-up with intensity 30% of MIP. The training will have 7 peaks of intensity with 70% of MIP for 60 sec, with 60-second of passive rest between the peaks, finishing the training with 20% of MIP for 2 min, totaling 17 min.
  Exercise: see group Combined aerobic/resistance exercise
  Interventions: Other: High-intensity IMT + Aerobic/resistance exercise
- Low-intensity IMT (Active Comparator): Low-intensity IMT + Aerobic/resistance exercise
  IMT:Training loads will be also adjusted weekly to the maximal inspiratory pressure (MIP). In the first two weeks as adaptation, the protocol will be of 2 minutes warm-up with intensity 20% of MIP. The training will be held with 3 sets of 15 repetitions, with 40% of MIP, finishing the training with 20% of MIP for 2 minutes. From the third week the protocol will be of 2 minutes warm-up with intensity 30% of MIP. The training will be held with 3 sets of 15 repetitions, with 60% of MIP, finishing the training with 30% of MIP for 2 minutes.
  Exercise: see group Combined aerobic/resistance exercise
  Interventions: Other: Low-intensity IMT + Aerobic/resistance exercise
- Aerobic/resistance exercise (Sham Comparator): Sham IMT + Aerobic/resistance exercise
  Aerobic session will consist of a 4-min of warm-up, 20 minutes of exercise, and 4 min of cool-down. Intensity will set by the formula: Training HR = (maximum HR - resting HR) × intensity % + resting HR. Patients will exercise using 30 seconds, high-intensity work phases 0.7% followed by 1-minute recovery bouts 0.5%. Resistance exercise will consist of dynamic lower and upper limb exercise. Upper limb exercises will include 3 sets of exercises for each muscle group performed with 10 repetitions each. Lower limb exercises will include 3 sets of exercises for each muscle group performed with 12 repetitions each. Resistance exercises will be performed at 12-MR.
  Interventions: Other: Sham IMT + Aerobic/resistance exercise

INTERVENTIONS:
Other: High-intensity IMT + Aerobic/resistance exercise — High-intensity IMT
  Arms: High-intensity IMT
Other: Low-intensity IMT + Aerobic/resistance exercise — Low-intensity IMT
  Arms: Low-intensity IMT
Other: Sham IMT + Aerobic/resistance exercise — Aerobic and resistance exercise
  Arms: Aerobic/resistance exercise

SUMMARY:
It is well-known that muscle weakness and deconditioning play an important role in low exercise capacity of patients with HF. Interestingly, not only peripheral muscles are impaired, but also respiratory muscles. Studies have shown that patients with HF may have, in addition to decreasing maximal inspiratory muscle strength and endurance, metabolic and structural impairments in diaphragm fibers. Moreover, exercise capacity and weakness of inspiratory muscles have been associated with low quality of life and poor prognosis, which make the addition of inspiratory muscle training (IMT) reasonable in cardiovascular rehabilitation.The specifications of the loads to be imposed during IMT is the main factor determining the outcome. Studies of IMT have highlighted the need for a fixed inspiratory workload during exercise. Thus, purpose of this report was to perform a randomized clinical trial of the effects of addition of high-intensity vs. low-intensity IMT to combined aerobic and resistance Exercise in patients with heart failure.

ELIGIBILITY:
Inclusion Criteria:

* The target population consists of adults patients aged ≥ 18 years with heart failure and New York Heart Association (NYHA) class I-III.

Exclusion Criteria:

* Unstable angina;
* coronary revascularization;
* Decompensated heart failure functional class IV (NYHA);
* Recent transplant or hospitalization (6 months <);
* Chronic Obstructive Pulmonary Disease;
* Neuromuscular, Orthopedic, Neurologic and Neoplastic Diseases;
* Recent myocardial infarction or cardiac surgery (less than 6 months);
* Atrial Fibrillation.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2017-08-01 (Actual); Primary Completion 2019-08-01 (Estimated); Study Completion 2020-08-01 (Estimated)

PRIMARY OUTCOMES:
Aerobic Capacity | 10 weeks
  Six-minute walk test
Health-Related Quality of Life: MLHFQ | 10 weeks
  Health-Related Quality of Life will be measured by a questionnaire (Minnesota Living with Heart Failure questionnaire - MLHFQ)

SECONDARY OUTCOMES:
Respiratory muscle strength | 10 weeks
  Maximal respiratory pressures
Disability | 10 weeks
  The World Health Organization Disability Assessment Schedule (WHODAS 2.0)

CONTACTS AND LOCATIONS:
Overall Officials: Mansueto Gomes-Neto, PhD, Principal Investigator — Federal University of Bahia
Locations (1):
- Mansueto Gomes Neto, Salvador, Estado de Bahia, Brazil